CLINICAL TRIAL: NCT05918861
Title: Phase III, Double-blind, Randomized Placebo-controlled Study to Evaluate the Effects of Dalcetrapib on Cardiovascular (CV) Risk in a Genetically Defined Population With a Recent Acute Coronary Syndrome (ACS)
Brief Title: Effect of Dalcetrapib on CV Risk in a Genetically Defined Population With a Recent ACS
Acronym: dal-GenE-2
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: DalCor Pharmaceuticals (Industry)
Collaborators: The Montreal Health Innovations Coordinating Center (MHICC) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DAL-302
Record Dates: First submitted 2023-06-15; First posted 2023-06-26 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Acute Coronary Syndrome
MeSH Terms: conditions — Acute Coronary Syndrome | interventions — dalcetrapib

STUDY DESIGN:
Intervention Model Description: Placebo-controlled, randomized, double-blind, parallel group, multi-center
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: With the exception of the statistician to the DSMB and the DSMB all other individuals will remain blinded until the final analysis of the primary study parameter.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dalcetrapib (Experimental): Dalcetrapib 600 mg (two 300 mg tablets) orally once daily
  Interventions: Drug: Dalcetrapib
- Placebo (Placebo Comparator): Matching dalcetrapib placebo tablets (2 tablets) orally once per day
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dalcetrapib — Cholesterol Ester Transfer Protein Inhibitor, 300 mg tablets
  Other Names: Cholesterol Ester Transfer Protein Inhibitor
  Arms: Dalcetrapib
Drug: Placebo — matching placebo tablets
  Other Names: Dalcetrapib matching placebo tablets
  Arms: Placebo

SUMMARY:
This is a placebo-controlled, randomized, double-blind, parallel group, phase 3 multicenter study in subjects recently hospitalized for ACS and with the appropriate genetic profile. Subjects will provide informed consent before any study-specific procedures are performed. A separate informed consent will be allowed for an initial pre-screening genetic testing. Subjects meeting the AA genotype will then consent to the full study and confirmatory genetic testing as required. Subject enrollment may begin in the hospital and will continue following release from the hospital or may begin following release from hospital. Screening procedures may be performed at the time of the index ACS event or anytime thereafter, with the condition that randomization must occur within the mandated window (up to12 weeks after the index event). Subjects will be assessed based on their medical history. Those who are likely to qualify will undergo Genotype Assay testing to evaluate genetic determination for the presence of AA genotype.

DETAILED DESCRIPTION:
This is an event-driven study and will last until approximately 200 subjects have experienced a primary event, unless the study is stopped at the planned interim analysis. Visits after randomization will be performed as virtual visits where permissible every 3 months or as clinic visits until the study is stopped. For any subject prematurely discontinuing study medication, assessments will be conducted every 3 months for the collection of study endpoints.

Those who are likely to qualify will undergo Genotype Assay Testing to evaluate genetic determination or the presence of the AA genotype at variant rs 1967309 in the ADCY9 gene as determined by the investigational use only version of the cobas ADCY9 Genotype Test, conducted at a designated investigational testing site.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with the appropriate genetic background and recently hospitalized for ACS (up to 3 months following the index event), will be enrolled in this trial.
* Both male and female subjects age 45 years and over at screening visit (V1)
* AA genotype at variant gene as determined by Genotype Assay Test, conducted at a designated investigational testing site (ITS)
* Clinically stable, ie, free of ischemic symptoms at rest or with minimal exertion for at least 1 week prior to randomization
* Prior to randomization, subjects must have evidence of guidelines-based management of LDL-C, at a minimum to include medical and dietary treatment.
* Randomization within 3 months of the index ACS event

Exclusion Criteria:

* Females who are pregnant (negative urine pregnancy test required for all women of child-bearing potential at Visit 2, Day 0) or breast-feeding
* Women of childbearing potential (women who are not surgically sterile or postmenopausal defined as amenorrhea for >12 months) who are not using at least one highly effective method of contraception.
* New York Heart Association (NYHA) Class III or IV heart failure
* Index ACS event presumed due to uncontrolled hypertension
* Systolic blood pressure (BP) >180 mmHg and/or diastolic blood pressure >110 mmHg at the time of randomization despite anti-hypertensive therapy
* Subjects with clinically apparent liver disease, eg, jaundice, cholestasis, hepatic synthetic impairment, active hepatitis or last known ALT or AST level >3 x ULN within 6 months prior to randomization (excluding index event)
* History of persistent and unexplained creatine phosphokinase (CPK) levels > 5 times the ULN as assessed within 6 months prior to randomization (excluding index event)
* Last known eGFR < 30 mL/min/1.73m2 as assessed within 6 months prior to randomization
* History of malignancy or any other significant comorbidity, the prognosis or management of which is likely to interfere with study conduct or subjects with a life expectancy of less than 3 years.
* Presence of any last known laboratory value as evaluated prior to randomization that is considered by the investigator to potentially limit the patient's successful participation in the study
* Subjects who have received any investigational drug within 1 month of randomization, or who expect to participate in any other investigational drug or device study during the conduct of this trial
* Subjects who have undergone coronary artery bypass graft (CABG) surgery between the index event and randomization

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2000 (Estimated)
Dates: Start 2023-10-03 (Actual); Primary Completion 2027-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Time to first occurrence of any fatal or non-fatal myocardial infarction (MI) | Average of 30 months from randomization
  Time to patients experiencing major cardiovascular events

SECONDARY OUTCOMES:
The composite of all-cause death, resuscitated cardiac arrest, non-fatal MI and non-fatal stroke | Average of 30 months from randomization
  Time to patients experiencing major cardiovascular events
Composite of all-cause death, resuscitated cardiac arrest, non-fatal MI and non-fatal stroke | Average of 30 months from randomization
  Time to patients experiencing first and recurrent occurrences
Fatal and non-fatal MI | Average of 30 months from randomization
  Time to patients experiencing first and recurrent occurrences

CONTACTS AND LOCATIONS:
Overall Officials: David Kallend, MBBS, Study Director — DalCor
Locations (194):
- United States (157):
  - Research Site, Alexander City, Alabama
  - Research Site, Birmingham, Alabama
  - Research Site, Fairhope, Alabama
  - Research Site, Huntsville, Alabama
  - Research Site, Mobile, Alabama
  - Research Site, Scottsdale, Arizona
  - Research Site, Tucson, Arizona
  - Research Site, Jonesboro, Arkansas
  - Research Site, North Little Rock, Arkansas
  - Research Site, Garden Grove, California
  - Research Site, Huntington Beach, California
  - Research Site, La Jolla, California
  - Research Site, Long Beach, California
  - Research Site, Los Angeles, California
  - Research Site, Newport Beach, California
  - Research Site, San Francisco, California
  - Research Site, Santa Barbara, California
  - Research Site, Stanford, California
  - Research Site, Torrance, California
  - Research Site, West Hills, California
  - Research Site, Aurora, Colorado
  - Research Site, Golden, Colorado
  - Research Site, Hartford, Connecticut
  - Research Site, New Haven, Connecticut
  - Research Site, Newark, Delaware
  - Research Site, Washington D.C., District of Columbia
  - Research Site, Boca Raton, Florida
  - Research Site, Clearwater, Florida
  - Research Site, Doral, Florida
  - Research Site, Fort Lauderdale, Florida
  - Research Site, Fort Myers, Florida
  - Research Site, Gainesville, Florida
  - Research Site, Hialeah, Florida
  - Research Site, Homestead, Florida
  - Research Site, Jacksonville, Florida
  - Research Site, Kissimmee, Florida
  - Research Site, Largo, Florida
  - Research Site, Miami, Florida
  - Research Site, Miami Lakes, Florida
  - Research Site, Ocala, Florida
  - Research Site, Pembroke Pines, Florida
  - Research Site, Pensacola, Florida
  - Research Site, Port Charlotte, Florida
  - Research Site, Safety Harbor, Florida
  - Research Site, Sarasota, Florida
  - Research Site, Tallahassee, Florida
  - Research Site, Tampa, Florida
  - Research Site, Winter Haven, Florida
  - Research Site, Acworth, Georgia
  - Research Site, Atlanta, Georgia
  - Research Site, Augusta, Georgia
  - Research Site, Gainesville, Georgia
  - Research Site, McDonough, Georgia
  - Research Site, Arlington Heights, Illinois
  - Research Site, Bloomingdale, Illinois
  - Research Site, Chicago, Illinois
  - Research Site, Glenview, Illinois
  - Research Site, Hazel Crest, Illinois
  - Research Site, Park Ridge, Illinois
  - Research Site, Springfield, Illinois
  - Research Site, Fort Wayne, Indiana
  - Research Site, Indianapolis, Indiana
  - Research Site, Merrillville, Indiana
  - Research Site, Munster, Indiana
  - Research Site, Newburgh, Indiana
  - Research Site, Richmond, Indiana
  - Research Site, Davenport, Iowa
  - Research Site, Iowa City, Iowa
  - Research Site, West Des Moines, Iowa
  - Research Site, Kansas City, Kansas
  - Research Site, Edgewood, Kentucky
  - Research Site, Lexington, Kentucky
  - Research Site, Louisville, Kentucky
  - Research Site, Hammond, Louisiana
  - Research Site, Lafayette, Louisiana
  - Research Site, Mandeville, Louisiana
  - Research Site, New Orleans, Louisiana
  - Research Site, Bangor, Maine
  - Research Site, Baltimore, Maryland
  - Research Site, Bethesda, Maryland
  - Research Site, Bowie, Maryland
  - Research Site, Columbia, Maryland
  - Research Site, Nottingham, Maryland
  - Research Site, Bay City, Michigan
  - Research Site, Dearborn, Michigan
  - Research Site, Detroit, Michigan
  - Research Site, Kalamazoo, Michigan
  - Research Site, Midland, Michigan
  - Research Site, Mount Clemens, Michigan
  - Research Site, Petoskey, Michigan
  - Research Site, Traverse City, Michigan
  - Research Site, Ypsilanti, Michigan
  - Research Site, Coon Rapids, Minnesota
  - Research Site, Duluth, Minnesota
  - Research Site, Minneapolis, Minnesota
  - Research Site, Saint Cloud, Minnesota
  - Research Site, Tupelo, Mississippi
  - Research Site, Springfield, Missouri
  - Research Site, St Louis, Missouri
  - Research Site, Lincoln, Nebraska
  - Research Site, Omaha, Nebraska
  - Research Site, Las Vegas, Nevada
  - Research Site, Bridgewater, New Jersey
  - Research Site, Hackensack, New Jersey
  - Research Site, Pomona, New Jersey
  - Research Site, Albuquerque, New Mexico
  - Research Site, Albany, New York
  - Research Site, Buffalo, New York
  - Research Site, Johnson City, New York
  - Research Site, New York, New York
  - Research Site, Poughkeepsie, New York
  - Research Site, Staten Island, New York
  - Research Site, Stony Brook, New York
  - Research Site, The Bronx, New York
  - Research Site, Pinehurst, North Carolina
  - Research Site, Rocky Mount, North Carolina
  - Research Site, Sanford, North Carolina
  - Research Site, Winston-Salem, North Carolina
  - Research Site, Canton, Ohio
  - Research Site, Cincinnati, Ohio
  - Research Site, Cleveland, Ohio
  - Research Site, Springfield, Ohio
  - Research Site, Toledo, Ohio
  - Research Site, Allentown, Pennsylvania
  - Research Site, Chambersburg, Pennsylvania
  - Research Site, Hershey, Pennsylvania
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, West Reading, Pennsylvania
  - Research Site, Wyomissing, Pennsylvania
  - Research Site, Providence, Rhode Island
  - Research Site, Rock Hill, South Carolina
  - Research Site, Spartanburg, South Carolina
  - Research Site, Rapid City, South Dakota
  - Research Site, Chattanooga, Tennessee
  - Research Site, Greeneville, Tennessee
  - Research Site, Jefferson City, Tennessee
  - Research Site, Memphis, Tennessee
  - Research Site, Oak Ridge, Tennessee
  - Research Site, Powell, Tennessee
  - Research Site, Amarillo, Texas
  - Research Site, Beaumont, Texas
  - Research Site, Corpus Christi, Texas
  - Research Site, Cypress, Texas
  - Research Site, Dallas, Texas
  - Research Site, Houston, Texas
  - Research Site, Kingwood, Texas
  - Research Site, McKinney, Texas
  - Research Site, Mesquite, Texas
  - Research Site, Port Arthur, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Victoria, Texas
  - Research Site, Waco, Texas
  - Research Site, Newport News, Virginia
  - Research Site, Norfolk, Virginia
  - Research Site, Richmond, Virginia
  - Research Site, Winchester, Virginia
  - Research Site, Seattle, Washington
- Canada (35):
  - Research Site, Calgary, Alberta
  - Research Site, Edmonton, Alberta
  - Research Site, Abbotsford, British Columbia
  - Research Site, Burnaby, British Columbia
  - Research Site, Kamloops, British Columbia
  - Research Site, North Vancouver, British Columbia
  - Research Site, Vancouver, British Columbia
  - Research Site, Victoria, British Columbia
  - Research Site, Winnipeg, Manitoba
  - Research Site, Moncton, New Brunswick
  - Research Site, St. John's, Newfoundland and Labrador
  - Research Site, Halifax, Nova Scotia
  - Research Site, Brampton, Ontario
  - Research Site, Cambridge, Ontario
  - Research Site, Kingston, Ontario
  - Research Site, London, Ontario
  - Research Site, Newmarket, Ontario
  - Research Site, Ottawa, Ontario
  - Research Site, Scarborough Village, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Chicoutimi, Quebec
  - Research Site, Granby, Quebec
  - Research Site, Greenfield Park, Quebec
  - Research Site, Laval, Quebec
  - Research Site, Lévis, Quebec
  - Research Site, Montreal, Quebec
  - Research Site, Québec, Quebec
  - Research Site, Rimouski, Quebec
  - Research Site, Saint-Charles-Borromée, Quebec
  - Research Site, Saint-Hubert, Quebec
  - Research Site, Saint-Jérôme, Quebec
  - Research Site, Terrebonne, Quebec
  - Research Site, Trois-Rivières, Quebec
  - Research Site, Sherbrooke, Quebec City
  - Research Site, Saskatoon, Saskatchewan
- Puerto Rico (2):
  - Research Site, Caguas, Puerto Rico
  - Research Site, Carolina

IPD SHARING:
Plan to Share IPD: No